CLINICAL TRIAL: NCT00840112
Title: Vitamin E Treatment for LCHAD Associated Neuropathy
Brief Title: Vitamin E Treatment for Long-Chain 3-Hydroxyacyl Coenzyme A (CoA) Dehydrogenase (LCHAD) Associated Neuropathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: New data does not support a role of vitamin E in LCHAD associated neuropathy.
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Oregon State University (Other)
Responsible Party: Melanie Gillingham, Ph.D., Oregon Health and Sciences University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OHSU eirb# 4929; F32DK065400 (NIH)
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2010-07

CONDITIONS: Peripheral Neuropathy; Mitochondrial Trifunctional Protein Deficiency
Keywords: Long-chain 3-hydroxyacyl CoA dehydrogenase (LCHAD); Mitochondrial trifunctional protein (TFP); LCHAD/TFP deficiency with peripheral neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases; Trifunctional Protein Deficiency With Myopathy And Neuropathy | interventions — alpha-Tocopherol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LCHAD/TFP with peripheral neuropathy (Experimental): Subjects diagnosed with LCHAD or TFP and with documented peripheral neuropathy
  Interventions: Dietary Supplement: Vitamin E supplement

INTERVENTIONS:
Dietary Supplement: Vitamin E supplement — 400 IU (268 mg) capsules of will be provided for the subjects. Subjects will be instructed to take one capsule with meals 2 times per day.
  Other Names: alpha tocopherol

SUMMARY:
Purpose:

People with a genetic defect in the ability to burn fat can also develop a problem with the nerves in their feet. The nerve problem, or neuropathy, can limit their ability to walk. Part of the treatment of their genetic defect in the ability to burn fat is to eat a very low fat diet. Vitamin E is found only in fatty foods like oils and nuts. People with a genetic defect in the ability to burn fat may have low vitamin E because of their low fat diet. The purpose of this study is to test whether vitamin E supplements can improve the nerve function in the feet of people with a genetic defect in the ability to burn fat.

Procedures:

Blood samples will be drawn at the beginning of the study, after 2 months and after 6 months of vitamin E supplements. The blood will be analyzed for plasma vitamin E concentrations. Around the time of each blood draw subjects will record all the food and beverages he or she consumes for three days. The subject will send the record to the investigator. Subjects will have a physical exam by a doctor specializing in nerves, a neurologist before and after taking vitamin E. They will have nerve function measured with a test called a nerve conduction velocity or NCV. Subjects will be given 800 international units (IU) of vitamin E per day for 6 months.

DETAILED DESCRIPTION:
People with long-chain 3-hydroxyacyl CoA dehydrogenase (LCHAD) or mitochondrial trifunctional protein (TFP) deficiency, inherited disorders of fatty acid ß-oxidation, lack an ability to fully oxidize fatty acids for energy. Progressive peripheral neuropathy is a chronic complication of these disorders that can lead to loss of the ability to walk in about 1/3 of the subjects. Current therapy for people with these disorders is based on frequent meals and consuming a low fat, very high carbohydrate diet. Severe restriction of dietary fat may lead to an iatrogenic fat-soluble vitamin deficiency. Vitamin E is a fat-soluble vitamin found in cooking oils, salad dressings, and nuts. Deficiency of vitamin E can result in a peripheral neuropathy similar to that described in subjects with LCHAD and TFP deficiency.

Hypothesis: Subjects with LCHAD or TFP deficiency are vitamin E deficient due to following a very low fat diet. Vitamin E deficiency exacerbates the peripheral neuropathy observed in this disease. High dose vitamin E supplementation will replete the vitamin E deficiency and improve neurological function in subjects with LCHAD or TFP deficiency.

Aim: Measure vitamin E concentrations and neurological function at baseline in 10 subjects with LCHAD or TFP deficiency. Following baseline measures, all subjects will be supplemented with high dose vitamin E (400 IU capsules 2 times per day) for 6 months. Vitamin E concentrations and neurological function studies will be repeated at the end of 6 months. Data from before and after vitamin E supplementation will be compared by students T-test.

Vitamin E functions as an antioxidant and has been used in multiple large supplementation trials. The upper limit of intake recommended as safe by the Institute of Medicine (IOM) is 600 mg or approximately 900 IU of vitamin E for children 9-13 years of age. We previously reported dietary intake of this vitamin was extremely low in children with LCHAD and TFP deficiency and should be supplemented (5). An iatrogenic vitamin E deficiency may exacerbate and/or accelerate neuropathic symptoms in subjects with LCHAD or TFP deficiency. This open-label trial tests the hypothesis that high dose vitamin E will improve neurological function in subjects with LCHAD and TFP deficiency who have progressive peripheral neuropathy.

Research Design and Methods:

Overall study design: This is an open-label supplementation trial of vitamin E in subjects with LCHAD or TFP deficiency. Subjects diagnosed with LCHAD or TFP and with documented peripheral neuropathy will be recruited to participate. A fasting baseline blood sample will be analyzed for plasma vitamin E concentrations. A neurological exam and nerve conduction studies (NCV) will be performed by a neurologist as a baseline measure of neuropathy. Subjects will begin high dose vitamin E supplementation for 6 months. 400 IU (268 mg) capsules of will be provided for the subjects. Subjects will be instructed to take one capsule with meals 2 times per day. The supplement is absorbed better when consumed with some fat from food. At the end of the 2 months of supplementation, another blood sample will be collected and analyzed for plasma vitamin E concentrations. At the end of 6 months, a 3rd blood sample will be collected and the neurological studies repeated. Differences in function and NCV from baseline will be correlated with plasma vitamin E concentrations. During the 6 months subjects will complete 2 3-day diet records to estimate vitamin E consumption from foods.

Blood Measures: Subjects will arrive to the clinic or lab for blood sampling after an overnight fast of a minimum of 8 hours but not more than 12 hours. Greater than 12 hours of fasting is not recommended for subjects with a fatty acid oxidation disorder. Six milliliters of venous whole blood will be collected . Plasma will be separated and frozen until analysis. Samples will be given a unique code in the laboratory of the principal investigator and shipped to Dr. Traber's laboratory in Corvallis, Oregon. Dr. Traber, at Oregon State University, will measure plasma vitamin E and vitamin E metabolites. The principal investigator will maintain the code to link data to patient information. Results from Dr. Traber's lab will be reported back to the principal investigator for data analysis.

Neurological Studies: A standard neurological examination will be carried out with an emphasis on the sensory exam, muscle weakness exam and deep tendon reflex exam. An electromyogram (EMG) and nerve conduction studies will also be carried out. For an EMG, a needle electrode is inserted through the skin into the muscle. The electrical activity detected by this electrode is displayed on an oscilloscope, and may be heard through a speaker. The observations of the wave forms by the physician will determine whether the electrical activity of the muscle is normal or whether pathological change such as denervation is present. Nerve conduction velocity (NCV) is a test of the speed of signals through a nerve. Patches called surface electrodes, similar to those used for ECG, are placed on the skin over the nerve at various locations. Each patch gives off a very mild electrical impulse, which stimulates the nerve. The nerve's resulting electrical activity is recorded by the other electrodes. The distance between electrodes and the time it takes for electrical impulses to travel between electrodes are used to determine the speed of the nerve signals. Further, the amplitude of the electrical discharge will be measured and the time that the impulse takes to cross the muscle-nerve junction will be determined. The electrical testing will involve both the motor and sensory nerves.

Statistical Analysis: Difference in plasma vitamin E concentrations and neurological studies between baseline and 6 months will be compared by student's T-test. Correlation between neurological outcomes and plasma vitamin E concentrations will be evaluated with linear regression.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of TFP, or LCHAD deficiency and progressive peripheral neuropathy
* Subjects must be > 7 years of age, and be willing to take vitamin E supplements.

Exclusion Criteria:

* None

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-07; Primary Completion 2015-07 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Plasma Vitamin E Concentrations | 6 months

SECONDARY OUTCOMES:
Neurological examinations: Sensory exam, muscle weakness exam and deep tendon reflex exam | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Gillingham, Ph.D, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Sciences University, Portland, Oregon, United States